CLINICAL TRIAL: NCT03009539
Title: Evaluating the Effectiveness of an eHealth EBI for Latino Youth in Primary Care
Brief Title: eHealth Evidence-based Intervention (EBI) for Latino Youth in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20160035; 1R01DA040756 (NIH)
Record Dates: First submitted 2016-11-29; First posted 2017-01-04 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Sexual Risk Behavior; Drug Use; Family Functioning
Keywords: Prevention with Hispanic youth; eHealth preventive intervention in primary care; Hispanic adolescent; Familias Unidas; eHealth Familias Unidas; effectiveness trial; sexually transmitted disease; parent-centered; Hispanic; sexual risk behavior
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Familias Unidas Primary Care (Experimental): eHealth Familias Unidas consists of 12 sessions: eight (12 - 15 minute) "mock" parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  Interventions: Behavioral: eHealth Familias Unidas Primary Care
- Treatment as Usual (No Intervention): Participants in this condition will not receive an intervention.

INTERVENTIONS:
Behavioral: eHealth Familias Unidas Primary Care — The experimental condition will consist of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
  Other Names: eHealth Familias Unidas
  Arms: eHealth Familias Unidas Primary Care

SUMMARY:
The purpose of this study is to test the relative effectiveness of a Hispanic-specific eHealth intervention, "e-Health Familias Unidas," in preventing and reducing drug use, sexual risk behaviors, and STIs among Hispanic youth in primary care. Families will be recruited through four pediatric primary care settings. Pediatric staff and research team members, including nurse assistants and mental health professionals, will implement eHealth Familias Unidas.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adolescents of Hispanic immigrant origin, defined by at least one parent born in a Spanish speaking country of the Americas. Parent must understand Spanish given that parent sessions are delivered in Spanish.
* Adolescent between the ages of 12 - 17 years
* Adolescent living with an adult primary caregiver who is willing to participate
* Families must have broadband internet access on a device, including (but not limited to) a smart phone, iPad, tablet, a home computer or a computer at another location (e.g., school, library, etc.)

Exclusion Criteria:

* Families reporting plans to move out of the South Florida area during the study period
* Families reporting that adolescent has been diagnosed with a developmental delay

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 921 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, Ph.D., Principal Investigator — University of Miami
Locations (12):
- United States (12):
  - PrimeCare Pediatrics, Hialeah, Florida
  - Ileana Fuentes Clinic, Miami, Florida
  - Ambulatory Care Center West Pediatrics at Jackson Memorial Hospital, Miami, Florida
  - UM Pediatric Mobile Clinic, Miami, Florida
  - UM UHealth Pediatrics at the Professional Arts Center, Miami, Florida
  - Borinquean Medical Centers, Miami, Florida
  - Borinquen Medical Centers, Miami, Florida
  - Kidstown Pediatrics, Miami, Florida
  - Belkys Bravo Clinic, Miami, Florida
  - Castro Pediatrics, Miami, Florida
  - University of Miami UHealth Pediatrics at Kendall, Miami, Florida
  - S. Florida Pediatric Partners, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional arms were added to include parent enrollments.
Groups:
- eHealth Familias Unidas Primary Care-Adolescents: eHealth Familias Unidas consists of 12 sessions: eight (12 - 15 minute) "mock" parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  eHealth Familias Unidas Primary Care: The experimental condition will consist of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
- Treatment as Usual-Adolescents: Participants in this condition will not receive an intervention.
- eHealth Familias Unidas Primary Care-Parents: Number of parents enrolled in the study's experimental condition
- Treatment as Usual-Parents: Number of parents enrolled in the study's control condition
Period: Overall Study
Arm/Group | eHealth Familias Unidas Primary Care-Adolescents | Treatment as Usual-Adolescents | eHealth Familias Unidas Primary Care-Parents | Treatment as Usual-Parents
Started | 225 | 231 | 225 | 231
Completed | 93 | 118 | 93 | 118
Not Completed | 132 | 113 | 132 | 113
Not completed — Lost to Follow-up | 132 | 113 | 132 | 113

BASELINE CHARACTERISTICS:
Groups:
- eHealth Familias Unidas Primary Care - Adolescents; eHealth Familias Unidas Primary Care - Parent: eHealth Familias Unidas consisted of 12 sessions: eight (12 - 15 minute) parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  eHealth Familias Unidas Primary Care: The experimental condition consisted of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
- Treatment as Usual - Adolescents; Treatment as Usual - Parent: Participants in this condition did not receive an intervention.
- Total: Total of all reporting groups
Arm/Group | eHealth Familias Unidas Primary Care - Adolescents | Treatment as Usual - Adolescents | eHealth Familias Unidas Primary Care - Parent | Treatment as Usual - Parent | Total
Number analyzed (Participants) | 225 | 231 | 225 | 231 | 912
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.96 (1.35) | 13.84 (1.35) | 43.46 (6.75) | 42.99 (6.58) | 13.90 (1.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 119 | 209 | 218 | 668
  Male | 103 | 112 | 16 | 13 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 225 | 231 | 225 | 231 | 912
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Drug Use
Description: Change in drug use will be reported as the episodes of reported drug use for the previous 90 days with questions from Monitoring the Future
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Population: The number of participants represent dyads. However, drug use was not analyzed for parents, only for adolescents. Therefore, these analyses include adolescents only.
Measure: Mean (Standard Deviation); unit: Episodes of drug use
Groups:
- eHealth Familias Unidas Primary Care: eHealth Familias Unidas Primary Care consists of 12 sessions: eight (12 - 15 minute) "mock" parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  eHealth Familias Unidas Primary Care: The experimental condition consisted of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
- Treatment as Usual: Participants in this condition did not receive an intervention.
Arm/Group | eHealth Familias Unidas Primary Care | Treatment as Usual
Number analyzed (Participants) | 225 | 231
Episodes of drug use
  Baseline | .02 (.22) | .50 (4.33)
  6 months post baseline | .09 (.69) | .34 (3.60)
  12 months post baseline | .07 (.58) | .59 (4.16)
  24 months post baseline | .12 (.73) | 1.46 (9.03)
  36 months post baseline | .22 (1.78) | 1.09 (8.11)

2. Primary Outcome: Change in Unprotected Sexual Behavior
Description: Change in unprotected sexual behavior was reported as endorsement incidence of having had sex without a condom during the previous 90 days using the Sexual Behavior Instrument. Higher values indicate worst outcomes.
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Population: The number of participants represent dyads. However, unprotected sexual behavior was not analyzed for parents, only for adolescents. Therefore, these analyses include adolescents only.
Measure: Mean (Standard Deviation); unit: Episodes of unprotected sexual behavior
Groups:
- eHealth Familias Unidas Primary Care: eHealth Familias Unidas consists of 12 sessions: eight (12 - 15 minute) "mock" parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  eHealth Familias Unidas Primary Care: The experimental condition consisted of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
Arm/Group | eHealth Familias Unidas Primary Care | Treatment as Usual
Number analyzed (Participants) | 225 | 231
Episodes of unprotected sexual behavior
  Baseline | .04 (.39) | .08 (.50)
  6 months post baseline | .04 (.33) | .08 (.50)
  12 months post baseline | .05 (.43) | .09 (.56)
  24 months post baseline | .13 (.66) | .19 (.78)
  36 months post baseline | .28 (.89) | .21 (.81)

3. Primary Outcome: Change in Incidence of Sexually Transmitted Infection
Description: Sexually transmitted infection incidence (i.e., gonorrhea and chlamydia) will be analyzed via a Polymerase Chain Reaction (PCR) from urine specimens
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Population: Analysis for the incidence of sexually transmitted infection was not conducted because the data were not collected. The data were not collected because we discontinued urine collection early on due to the COVID pandemic and associated shutdowns.
Arm/Group | eHealth Familias Unidas Primary Care | Treatment as Usual
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Family Functioning as Assessed by the Parenting Practices Questionnaire
Description: Change in family functioning will be reported using the Parenting Practices Scale (Tolan et al., 1997). Subscales include positive parenting (9 items, alpha = .78 for adolescents; alpha = .77 for parents) parental involvement( 20 items, alpha = .86 for adolescents; alpha = .85 parents). Responses range from 0 to 4 with higher values indicating better parenting, higher scores indicate more positive outcomes. The mean for each subscale was used to create a sum score.
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- eHealth Familias Unidas Primary Care-Parent; eHealth Familias Unidas Primary Care-Adolescent: eHealth Familias Unidas consists of 12 sessions: eight (12 - 15 minute) "mock" parent sessions in Spanish and four (30 - 45 minute) online family sessions delivered in either Spanish and/or English.
  eHealth Familias Unidas Primary Care: The experimental condition consisted of "eHealth Familias Unidas Primary Care." eHealth Familias Unidas Primary Care is an adaptation of the face-to-face version of Familias Unidas. As with face-to-face Familias Unidas, eHealth Familias Unidas Primary Care aims to prevent drug use, sexual risk behaviors, and STIs by improving family functioning. Similar to face-to-face Familias Unidas, eHealth Familias Unidas is a multi-level intervention that targets risk and protective factors at the multiple systems affecting the youth and youths' family.
- Treatment as Usual-Parent; Treatment as Usual-Adolescent: Participants in this condition did not receive an intervention.
Arm/Group | eHealth Familias Unidas Primary Care-Parent | Treatment as Usual-Parent | eHealth Familias Unidas Primary Care-Adolescent | Treatment as Usual-Adolescent
Number analyzed (Participants) | 225 | 231 | 225 | 231
score on a scale
  Baseline positive parenting | 23.66 (4.9) | 24.08 (4.85) | 21.9 (6.02) | 22.64 (6.54)
  6 month positive parenting | 23.83 (4.75) | 23.45 (5.0) | 22.10 (6.02) | 22.10 (5.88)
  12 month positive parenting | 23.85 (4.72) | 23.32 (4.67) | 22.09 (5.98) | 22.36 (6.05)
  24 months positive parenting | 23.71 (4.73) | 23.26 (5.27) | 21.78 (6.42) | 21.67 (6.38)
  36 month positive parenting | 22.50 (5.17) | 22.81 (4.92) | 21.89 (6.46) | 22.17 (6.56)
  baseline parental involvement | 50.49 (8.40) | 51.60 (7.94) | 41.98 (9.60) | 42.19 (9.23)
  6 month parental involvement | 50.66 (7.93) | 50.54 (7.54) | 41.62 (9.01) | 41.62 (9.30)
  12 month parental involvement | 50.71 (8.53) | 50.24 (8.40) | 41.81 (9.16) | 41.35 (8.90)
  24 month parental involvement | 49.58 (8.96) | 49.16 (8.76) | 40.90 (10.17) | 40.17 (9.88)
  36 month parental involvement | 48.43 (9.64) | 48.02 (9.01) | 40.58 (10.35) | 40.34 (10.44)

5. Secondary Outcome: Change in Family Functioning as Assessed by the Parent Relationship With Peer Group
Description: Change in family functioning will be reported using the Parent Relationship with Peer Group. The Parent Relationship with Peer Group is a six item measure with response items ranging from 0 to 24. Higher scores indicate better outcomes.The mean was used to create a sum score.
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eHealth Familias Unidas Primary Care-Parent | Treatment as Usual-Parent | eHealth Familias Unidas Primary Care-Adolescent | Treatment as Usual-Adolescent
Number analyzed (Participants) | 225 | 231 | 225 | 231
score on a scale
  Baseline | 11.90 (4.2) | 11.67 (4.49) | 9.67 (4.6) | 9.42 (4.46)
  6 months post baseline | 11.90 (4.33) | 11.87 (4.33) | 9.77 (4.36) | 8.93 (4.59)
  12 months post baseline | 11.92 (4.36) | 11.88 (4.09) | 9.56 (4.70) | 8.95 (4.85)
  24 months post baseline | 11.59 (4.26) | 11.78 (4.31) | 9.44 (4.63) | 8.96 (4.58)
  36 months post baseline | 11.25 (4.39) | 10.70 (4.3) | 9.06 (4.64) | 8.25 (4.67)

6. Secondary Outcome: Change in Family Functioning as Assessed by the Parent-Adolescent Communication Scale
Description: Change in family functioning will be reported using the Parent-Adolescent Communication Scale. The Parent-Adolescent Communication Scale is a twenty-item questionnaire with a total score ranging from 20 to 100 with higher scores indicating better communication.The mean was used to create a sum score.
Time Frame: Baseline, Baseline to 6 months, baseline to 12 months, baseline to 24 months, baseline to 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eHealth Familias Unidas Primary Care-Parent | Treatment as Usual-Parent | eHealth Familias Unidas Primary Care-Adolescent | Treatment as Usual-Adolescent
Number analyzed (Participants) | 225 | 231 | 225 | 231
score on a scale
  Baseline | 76.28 (9.92) | 76.29 (10.36) | 71.47 (13.61) | 71.67 (13.3)
  6 months post baseline | 77.55 (10.00) | 77.64 (10.44) | 72.87 (14.75) | 71.99 (15.01)
  12 months post baseline | 78.15 (9.44) | 77.10 (11.11) | 72.31 (13.21) | 71.39 (15.03)
  24 months post baseline | 79.85 (10.18) | 77.46 (11.95) | 71.66 (14.40) | 70.84 (15.04)
  36 months post baseline | 79.52 (10.74) | 77.70 (11.47) | 70.57 (16.27) | 69.63 (15.80)

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Adverse events were not monitored for caregivers.
Arm/Group | eHealth Familias Unidas Primary Care | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/231
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/231
Other Adverse Events (participants affected / at risk) | 0/225 | 0/231

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03009539/Prot_SAP_002.pdf
  • Informed Consent Form (2017-04-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03009539/ICF_003.pdf